CLINICAL TRIAL: NCT06388135
Title: Serplulimab Combined With Nab-paclitaxel and Cisplatin in Neoadjuvant Therapy for Resectable Esophageal Squamous Cell Carcinoma: a Study Protocol of Prospective Single-center, Open Label and Exploratory Cohort Study (SNC-01)
Brief Title: Serplulimab Combined With Nab-paclitaxel and Cisplatin in Neoadjuvant Therapy for Resectable Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yang Jianjun, PhD (Other)
Responsible Party: Sponsor-Investigator, Yang Jianjun, PhD, Professor from Xijing Hospital, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNC-01
Record Dates: First submitted 2024-04-18; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — 130-nm albumin-bound paclitaxel; Cisplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serplulimab，nab-paclitaxel，Cisplatin (Experimental): Serplulimab (200 mg), cisplatin (60-75 mg/m2), and nab-paclitaxel (135 mg/m2) administered intravenously at the beginning of every 3-week cycle
  Interventions: Drug: Serplulimab Combined With Nab-paclitaxel and Cisplatin
- nab-paclitaxel，Cisplatin (Sham Comparator): Cisplatin (60-75 mg/m2) and nab-paclitaxel (135 mg/m2) given intravenously at the beginning of every 3-week cycle.
  Interventions: Drug: nab-paclitaxel，Cisplatin

INTERVENTIONS:
Drug: Serplulimab Combined With Nab-paclitaxel and Cisplatin — Serplulimab (200 mg), cisplatin (60-75 mg/m2), and nab-paclitaxel (135 mg/m2) administered intravenously at the beginning of every 3-week cycle.
  Arms: Serplulimab，nab-paclitaxel，Cisplatin
Drug: nab-paclitaxel，Cisplatin — nab-paclitaxel，Cisplatin
  Arms: nab-paclitaxel，Cisplatin

SUMMARY:
Abstract Objective: This study aims to investigate the potential clinical impact of neoadjuvant immunotherapy in resectable esophageal squamous cell carcinoma (ESCC).

The efficacy and safety of combining the programmed death 1 (PD-1) inhibitor serplulimab with nab-paclitaxel and cisplatin as neoadjuvant therapy in patients with resectable ESCC will be evaluated. Methods and analysis: A prospective, single-center, open-label cohort study will enroll 80 patients, with 40 patients allocated to the experimental group and 40 patients to the control group. Patients in the experimental arm will undergo 3 cycles of neoadjuvant therapy comprising serplulimab, cisplatin, and nab-paclitaxel, while those in the control arm will receive 3 cycles of neoadjuvant therapy with cisplatin and nab-paclitaxel. The primary efficacy endpoint will be the assessment of pathological complete response (pCR) following neoadjuvant therapy. Secondary efficacy endpoints will include major pathological response (MPR), disease-free survival, objective response rate (ORR), and monitoring of adverse events (AEs).

Ethics: Ethics approval has been obtained from the Ethics Committee at the First Affiliated Hospital (Xijing Hospital) of Air force Military Medical University (KY20242052-C-1).

ELIGIBILITY:
Inclusion criteria:

* The age range of the enrolled patients was 18-70 years;
* ECOG score 0-1 ;
* Patients with ESCC diagnosed by pathology (histology or cytology);
* Resectable IB-III (cT1b~3N1-2M0 or cT3~4aN0~1M0) stage per the 8th edition of clinical TNM staging;
* Measurable lesions (per RECIST 1.1 criteria: major tumor diameter on CT scan ≥10mm, short lymph node diameter on CT scan ≥15mm);
* No prior radiotherapy, chemotherapy, surgery, or targeted therapy;
* Surgical tolerance and ability to consume liquid diet without esophageal complications;
* Normal major organ function criteria: (1) Blood tests: ANC ≥ 1.5 × 109/L, PLT ≥ 100 × 109/L, HB ≥ 90 g/L; (2) Biochemical tests: TBIL≤1.5×ULN, ALT/AST≤ 2.5×ULN, serum creatinine ≤1.5×ULN, ALB ≥ 30 g/L; (3) Coagulation function: INR≤1.5×ULN, APTT≤1.5×ULN;
* Normal or mildly to moderately abnormal lung function suitable for EC surgery: A) VC%>60%, B) FEV1>1.2L, FEV1%>40%, C) DLCO>40%;
* Voluntary participation with informed consent and good compliance.

The exclusion criteria were as follows:

* Any current or past presence of autoimmune diseases;
* Patients with immune deficiency disorders like HIV infection, active hepatitis B (HBV DNA ≥ 500 IU/ML), hepatitis C (HCV antibody positive, and HCV-RNA above the detection limit), or co-infection with hepatitis B and hepatitis C;
* Patients who have taken immunosuppressive drugs within 14 days before enrollment; patients who experienced a weight loss of ≥10% within 6 months prior to enrollment, or have a BMI below 18.5kg/m2, or have a PG-SGA score indicating grade C;
* Patients who had attenuated live vaccines within 4 weeks before enrollment;
* History of other cancers;
* Patients with myocardial infarction within six months before enrollment or diagnosed with New York Heart Association grade ≥ II heart failure;
* Patients who have experienced severe infections or undergone allogeneic organ transplantation or hematopoietic stem cell transplantation within the 4 weeks preceding enrollment;
* Patients with substance abuse, alcohol consumption, or psychotropic substance use.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
pCR | after surgery,within 12 weeks
  pathological Complete Response

SECONDARY OUTCOMES:
MPR | after surgery,within 12 weeks
  major pathologic response
DFS | up to 24 months
  Disease free survival
ORR | up to 24 months
  objective response rate
AEs | up to 24 months
  adverse events